CLINICAL TRIAL: NCT03109730
Title: A Phase 1b/2a, Dose-Ranging Study of the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of ABI-H0731 in Patients With Chronic Hepatitis B
Brief Title: Phase 1b/2a Study of ABI-H0731 in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ABI-H0731-101B
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cohort B1 (Experimental): ABI-H0731 or Placebo in varying doses by mouth for 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731
- Cohort B2 (Experimental): ABI-H0731 or Placebo in varying doses by mouth for 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731
- Cohort B3 (Experimental): ABI-H0731 or Placebo in varying doses by mouth for 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731
- Cohort B4 (Experimental): ABI-H0731 or Placebo in varying doses by mouth for 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731
- Cohort B5 (Experimental): ABI-H0731 or Placebo in combination with entecavir or tenofovir for 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731; Drug: Entecavir; Drug: Tenofovir Disoproxil Fumarate
- Cohort B6 (Experimental): ABI-H0731 or Placebo, in combination with a commerically-approved nucleos(t)ide plus PegIFN in treatment-experienced patients, for 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731; Drug: Pegasys

INTERVENTIONS:
Drug: ABI-H0731 — A novel HBV core protein allosteric modifier (CpAM) which is being developed as a potential therapeutic advance for CHB patients
Drug: Placebo for ABI-H0731 — Sugar pill manufactured to mimic the ABI-H0731 tablet
Drug: Entecavir — An antiviral medication used in the treatment of hepatitis B virus infection
  Other Names: ETV
  Arms: Cohort B5
Drug: Tenofovir Disoproxil Fumarate — An antiviral medication used in the treatment of hepatitis B virus infection
  Other Names: TDF
  Arms: Cohort B5
Drug: Pegasys — Used to treat adults with chronic hepatitis B virus who show signs of liver damage
  Other Names: peginterferon alfa-2a
  Arms: Cohort B6

SUMMARY:
The purpose of this protocol is to obtain pharmacodynamic and pharmacokinetic data on ABI-H0731 and to provide the opportunity for preliminary evaluation of combination therapy of ABI-H0731 with currently approved antiviral treatment for chronic hepatitis B.

DETAILED DESCRIPTION:
The Phase 1b/2a assessments of the dose-related safety, PK, and initial antiviral efficacy of ABI-H0731 in hepatitis B patients will be conducted at approximately 17 different sites to meet enrollment goals of 108 chronic hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age
* Chronic HBV infection
* Body Mass Index (BMI) 18-38 kg/m2 and a minimum body weight of 45 kg

Exclusion Criteria:

* Seropositive for HIV, HCV, or HDV antibody at Screen
* Previous treatment with any investigational HBV antiviral treatments within the last 6 months
* Other known cause of liver disease, including NASH
* Other medical condition that requires persistent medical management or chronic or recurrent pharmacologic or surgical intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with chronic HBV infection with treatment-related adverse events and laboratory abnormalities as assessed by CTCAE v4.0. | Up to 57 days

CONTACTS AND LOCATIONS:
Locations (14):
- Australia (4):
  - Monash University, Clayton, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- University of Hong Kong, Hong Kong, Hong Kong
- South Korea (4):
  - Hallym University, Chuncheon
  - CHA Bundang Medical Center, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Severance Hospital, Yonsei University, Seoul
- Taiwan (2):
  - Keelung Chang Gung Memorial Hospital, Keelung
  - National Taiwan University Hospital, Taipei
- United Kingdom (3):
  - King's College Hospital, London
  - Royal Free Hospital NHS Foundation Trust, London
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided